CLINICAL TRIAL: NCT04317677
Title: Effects of Bladder Voiding on Sleep Architecture in Infants
Acronym: MIDESOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0223
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Babies hospitalized in the pediatric sleep unit (Other)
  Interventions: Other: Study of the effect of bladder voiding on sleep fragmentation during day and night sleep

INTERVENTIONS:
Other: Study of the effect of bladder voiding on sleep fragmentation during day and night sleep — Vigilance state of babies will be continuously recorded during the first 24 hours of hospitalization by polysomnography and actigraphy. In parallel, bladder voiding episodes will be detected with an innovative device placed on babies diapers.

SUMMARY:
Sleep changes rapidly during the first year of life. Brain maturation is accompanied by sleep consolidation in several episode during day and night (daytime naps and night sleep) and progressive organization during the 24h period (more wake during day et more sleep during night). In the first months of life, sleep episodes are frequently interrupted by wake, possibly induced by multiple external and internal stimuli. One of this stimulus could be bladder voiding that is particularly frequent in babies. Only one team worked on the link between sleep and bladder voiding and reported that bladder voiding was associated with cortical arousal during a daytime nap in a little group of babies.

In this study, investigators propose to study the relationship between sleep and bladder voiding in a bigger group of infant and during daytime but also nighttime sleep.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both sex
* Age ≥1 month and ≤ 12 months
* Referred to the sleep unit for sleep trouble screening following ALTE (Apparent Life Threatening Event).
* Patients should benefit from appropriate insurance system
* Parents who have expressed a willingness to participate in the study, who have signed and dated the informed consent.

Exclusion Criteria:

* Neurological, endocrinal or syndromic diseases :

  * Head and neck congenital malformations
  * Pierre Robin Syndrome
  * Trisomy
  * Achondroplasia
  * Prader Willy syndrome
  * Ondine syndrome
  * Cardiac diseases and malformations
* Weight <2.5 kg
* Preterm babies (under 37 weeks of gestational age)

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of arousals / awakenings in a timely relation with bladder voiding. | 24 hours
  The occurrence of arousals and awakenings will be determined form polysomnography signals including electroencephalogram (EEG), electrooculogram (EOG) and a electromyogram (EMG). Arousals and awakenings will be scored as defined by the international rules for visual scoring of EEG (AASM manual 2007). Investigators will calculate the percentage of bladder voiding episode leading to arousal / awakening events

SECONDARY OUTCOMES:
Sleep stage following bladder voiding events | 24 hours
  Sleep stages will be scored as defined by the international rules (AASM 2007). Investigators will determine the proportion of bladder voiding events leading to a change of sleep stage.
EEG frequencies following bladder voiding episodes | 24 hours
  EEG will be quantitatively analyzed and the power spectrum in each frequency band will be determined. Investigators will determine the proportion of bladder voiding events followed by a significant change of EEG frequencies.
Heart rate following bladder voiding episode | 24 hours
  EKG will be obtained during the entire record. Investigators will determine the proportion of bladder voiding followed by a significant change of heart rate
Activity record with actigraphy in babies | 24 hours
  Coherence analysis between actigraphy and polysomnography records

CONTACTS AND LOCATIONS:
Locations (1):
- Service épilepsie, sommeil et explorations neuropédiatriques, Hôpital Femme mère enfant - Groupement hospitalier Est - HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No